CLINICAL TRIAL: NCT07233590
Title: The Effect of Apical Patency on Postoperative Pain Following Root Canal Treatment of Single-Rooted Teeth: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Apical Patency on Postoperative Pain Following Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Pricipal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10.05.2024/33
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain After Endodontic Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Patency Group (Active Comparator): Preoperative pain was recorded using a Numerical Rating Scale (NRS) before treatment. All procedures were performed in a single visit by one operator under 3× magnification. Local anesthesia was achieved with 4% articaine containing 1:100,000 epinephrine. After rubber dam isolation, caries and existing restorations were removed and an endodontic access cavity was prepared under copious water cooling using high-speed sterile diamond burs.
  The working length was established with an electronic apex locator (Root ZX Mini) and confirmed radiographically. In this group, apical patency was not maintained: after working length determination, all subsequent instrumentation was confined within the working length, and no file was advanced beyond the apical foramen.
  Root canals were shaped using the One Curve NiTi rotary system (25/.06 or 35/.04) with a crown-down technique. During shaping, canals were irrigated with a total of 10 mL of 2.5% sodium hypochlorite (2 mL after each shaping step) de
  Interventions: Procedure: Root canal treatment without apical patency
- Patency Group (Experimental): Preoperative pain was recorded using a Numerical Rating Scale (NRS) before treatment. All procedures were performed in a single visit by one operator under 3× magnification. Local anesthesia was achieved with 4% articaine containing 1:100,000 epinephrine. After rubber dam isolation, caries and existing restorations were removed and an endodontic access cavity was prepared under copious water cooling using high-speed sterile diamond burs.
  The working length was established with an electronic apex locator (Root ZX Mini) and confirmed radiographically. In this group, apical patency was maintained: a #10 K-file was gently advanced 1 mm beyond the working length at each instrument change to prevent apical blockage, remove accumulated debris, and facilitate irrigant delivery to the apical terminus.
  Root canals were shaped using the One Curve NiTi rotary system (25/.06 or 35/.04) with a crown-down technique. During shaping, canals were irrigated with a total of 10 mL of 2.5% sodium hypochl
  Interventions: Procedure: Root canal treatment with apical patency

INTERVENTIONS:
Procedure: Root canal treatment with apical patency — Single-visit root canal treatment of asymptomatic vital single-rooted teeth in which apical patency is maintained. After working length determination with an electronic apex locator and radiographic confirmation, a #10 K-file is gently extended 1 mm beyond the working length at each instrument change to prevent apical blockage, remove debris, and facilitate irrigant delivery to the apical terminus. All other steps, including anesthesia, rubber dam isolation, access cavity preparation, rotary shaping with the One Curve NiTi system, standardized irrigation with 2.5% NaOCl and 17% EDTA, obturation, and definitive composite restoration, follow a standardized protocol.
  Arms: Patency Group
Procedure: Root canal treatment without apical patency — Single-visit root canal treatment of asymptomatic vital single-rooted teeth in which apical patency is not maintained. After working length determination with an electronic apex locator and radiographic confirmation, all subsequent instrumentation is confined within the working length and no file is advanced beyond the apical foramen. All other steps, including anesthesia, rubber dam isolation, access cavity preparation, rotary shaping with the One Curve NiTi system, standardized irrigation with 2.5% NaOCl and 17% EDTA, obturation, and definitive composite restoration, follow the same standardized protocol as in the patency group.
  Arms: Non-Patency Group

SUMMARY:
The goal of this randomized controlled clinical trial was to evaluate whether implementing apical patency affects the intensity of postoperative pain after single-visit root canal treatment in asymptomatic, vital, single-rooted teeth.

The main question it aims to answer is:

Does maintaining apical patency by gently extending a #10 K-file 1 mm beyond the working length during canal shaping influence postoperative pain compared with instrumentation confined within the working length?

In the patency group, the working length was determined with an electronic apex locator and radiograph, and then apical patency was maintained by passively extending a #10 K-file 1 mm beyond the working length at each instrument change to prevent apical blockage, remove debris, and facilitate irrigant delivery to the apical terminus.

In the non-patency group, the working length was likewise established with an electronic apex locator and radiograph, but all subsequent instrumentation was confined within the working length and no file was advanced beyond the apical foramen.

In both groups, all other clinical procedures-including anesthesia, rubber dam isolation, access cavity preparation, rotary canal shaping with the One Curve NiTi system, standardized irrigation with 2.5% NaOCl and 17% EDTA, obturation with gutta-percha and epoxy resin-based sealer, and definitive composite restoration-were performed in a single visit using the same protocol. Postoperative pain was recorded on a Numerical Rating Scale (NRS) at 0-6, 6-12, 12-24, 24-36, and 36-48 hours, and analgesic intake within 48 hours was documented.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years, classified as ASA I or ASA II according to the American Society of Anesthesiologists (ASA), who had not taken analgesics for at least 6 hours prior to treatment.
* Asymptomatic, single-rooted vital teeth without spontaneous pain (including teeth perforated during prosthetic preparation or teeth adjacent to a cyst in an area scheduled for cyst surgery).
* Radiographic evidence of mature apices with no periapical pathology; periodontal probing depth ≤ 3 mm; and gingival health meeting Glickman's criteria.
* Individuals who are literate, able to provide written informed consent, and capable of understanding and using the pain scale.

Exclusion Criteria:

* Patients who are pregnant or have a cardiac pacemaker.
* Patients who used antibiotics within the past month or who required antibiotic prophylaxis.
* Presence of extensive restorations in the tooth of interest.
* Patients reporting concurrent pain in adjacent teeth.
* Dental or orofacial pain of non-endodontic origin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Up to 48 hours after treatment.
  The numerical rating scale for pain is an 11-point scale from 0 to 10, where 0 means no pain and 10 means the worst pain imaginable. The patient is asked to choose the number that best represents the intensity of pain he or she feels at that moment. It is used to assess the severity of postoperative pain and to help evaluate the need for and response to analgesic medication. Also called NRS.

CONTACTS AND LOCATIONS:
Overall Officials: Adile Şehnaz Yılmaz, DDS, Phd, Professor, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaylali IE, Demirci GK, Kurnaz S, Celik G, Kaya BU, Tunca YM. Does Maintaining Apical Patency during Instrumentation Increase Postoperative Pain or Flare-up Rate after Nonsurgical Root Canal Treatment? A Systematic Review of Randomized Controlled Trials. J Endod. 2018 Aug;44(8):1228-1236. doi: 10.1016/j.joen.2018.05.002. Epub 2018 Jun 20. PMID 29935875